CLINICAL TRIAL: NCT01865669
Title: In-vitro Myometrial Contractility After Oxytocin Pre-exposure in Women With Advanced Maternal Age and Morbid Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-04
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Postpartum Hemorrhage
Keywords: Uterine contraction; Dose response; Oxytocin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): A control sample from each patient (no oxytocin applied) will be measured concurrently with samples treated with varying concentrations of oxytocin.
- Oxytocin (Experimental): Samples from each patient will be bathed in a solution containing varying concentrations of oxytocin.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin, 10-10mol/L to 10-5mol/L
  Other Names: pitocin
  Arms: Oxytocin

SUMMARY:
Women with advanced maternal age and morbid obesity, have a higher incidence of labor induction/ augmentation and cesarean section (CS), and are at a greater risk for postpartum hemorrhage (PPH). Oxytocin is the first line drug in the treatment of PPH, however, oxytocin receptor (OTR) desensitization has been recognized in the context of prolonged labors secondary to either endogenous or exogenous oxytocin exposure. It is unknown if oxytocin desensitization specifically affects contractility in women with advanced maternal age and morbid obesity when compared to younger or normal weight populations. Further it is not known if the higher incidence of PPH seen in these women is due to poor uterine contractility and/or poor response to oxytocin.

The investigators hypothesize that women with advanced maternal age and morbid obesity will exhibit poor myometrial contractility as compared to women that are younger and of normal body habitus, in both oxytocin pre-treated and untreated myometrium.

DETAILED DESCRIPTION:
In view of the growing concern over the rising incidence of later maternal age and morbid obesity in the obstetric population, scientific evidence on pregnancy outcomes in these patients is timely and important. The investigators' previously validated in-vitro model provides a solid foundation for the study of myometrial contractility under controlled conditions, without any confounders that could be encountered in clinical settings. It is also likely to provide in-depth understanding of the parameters that the investigators feel are responsible for higher incidence of PPH in these patients. The investigators' study will form a basis for future modifications in oxytocin augmentation regimens and pharmacotherapy for control of PPH in these patient populations.

ELIGIBILITY:
Inclusion Criteria:

* patients who give written informed consent
* patients requiring elective primary or 1st repeat Cesarean section
* patients with gestational age 37-41 weeks
* non-labouring patients, not exposed to exogenous oxytocin
* Cesarean section under spinal anesthetic
* patients <30 years of age with a normal pre-pregnancy BMI (20 and 24.9 kg/m2)
* patients ≥40 years of age with a normal pre-pregnancy BMI
* patients with a BMI≥40 kg/m2 and age <30 years

Exclusion Criteria:

* patients who refuse to give written informed consent
* patients who require general anesthesia
* patients who have had more than one previous uterine surgery/CS
* patients with placental abnormalities (abruption, accreta, percreta)
* patients with bleeding disorders
* presence of any other risk factors for PPH

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-05; Primary Completion 2017-06-13 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
Motility index | 6-8 hours

SECONDARY OUTCOMES:
Amplitude of contraction | 6-8 hours
Integrated area under response curve (AUC) | 6-8 hours
Frequency of contraction | 6-8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luca AM, Carvalho JCA, Ramachandran N, Balki M. The effect of morbid obesity or advanced maternal age on oxytocin-induced myometrial contractions: an in vitro study. Can J Anaesth. 2020 Jul;67(7):836-846. doi: 10.1007/s12630-020-01615-6. Epub 2020 Mar 18. PMID 32189217